CLINICAL TRIAL: NCT02556060
Title: Lamotrigine for Ketamine Dependence: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Lamotrigine for Ketamine Dependence Trial
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Taipei City Hospital (Other Government)
Collaborators: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Lin, Shih-Ku, Chair of Department of Psychiatry, Taipei City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TCHIRB-102309
Record Dates: First submitted 2015-09-08; First posted 2015-09-22 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Addiction
Keywords: ketamine use disorder; lamotrigine; craving
MeSH Terms: conditions — Behavior, Addictive | interventions — Lamotrigine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lamotrigine (Experimental): lamotrigine extended release up to 200 mg/day,
  Interventions: Drug: Lamotrigine; Drug: Placebo
- Placebo (Placebo Comparator): Identical Placebo
  Interventions: Drug: Lamotrigine; Drug: Placebo

INTERVENTIONS:
Drug: Lamotrigine — Starting from 25 mg/day in the first week, then titrated up to 200 mg/day for 12 weeks
  Other Names: Lamofree ER
Drug: Placebo — Same dosing schedule as study drug
  Other Names: Identical to Lamofree ER

SUMMARY:
The purpose of this study is to investigate the efficacy of lamotrigine in the treatment of ketamine dependence in a double-blind, placebo controlled design.

DETAILED DESCRIPTION:
Introduction

Ketamine is an anesthetic derivative of phencyclidine (PCP; 'Angel dust') with dissociative, analgesic and psychedelic properties. Recreational use of ketamine was first documented on the west coast of the United States in the early 1970s. Ketamine is frequently described as a "unique drug" because it shows hypnotic (sleep producing), analgesic (pain relieving) and amnesic (short-term memory loss) effects; no other drug used in clinical practice combines these three important features at the same time. Ketamine produces an anaesthetic state, which has been termed "dissociative anaesthesia", characterized by analgesia and changes in vigilance and perception, but it is not a sedative or hypnotic. It appears that ketamine selectively interrupts the thalamocortical system. Ketamine has some anxiolytic- and antidepressant-like properties in sub-anesthetic doses.

Mechanism of ketamine addiction

The existence of binding sites for PCP and ketamine were first identified in 1979. Earlier reports indicate that ketamine essentially blocks the N-methyl-D-aspartate (NMDA) subtype of glutamate receptors. The antagonism of NMDA receptor is responsible for its specific properties including psychedelic, anesthetic, analgesic, anxiolytic, antidepressant, hypnotic effects and cognitive impairment. In fact, ketamine also binds to non-NMDA glutamate receptors and involves glutamate-independent mechanisms associated with nicotinic and muscarinic cholinergic, monoaminergic and opioid receptors.

Currently there is no specific pharmacological treatment model for ketamine dependence. Continuous urine screen plus medications for psychiatric symptoms treatment revealed fair results.

Study drug: Lamotrigine

Lamotrigine is an anticonvulsant drug used in the treatment of epilepsy and bipolar disorder. Besides it's sodium channels blocking effect as an antiepileptic drugs, lamotrigine also inhibits the release of glutamate through modulation of high voltage-activated calcium currents and sodium channels.

Method

Patient Patients with ketamine use disorder seeking treatment at Taipei City Hospital and Psychiatric Center will be invited to participate this clinical trial. Treatment and assessment Schedule After informed consent signature with explanations about the procedure of this study, the initiation includes collecting drug use history and medical history, conducting a physical examination, and performing clinical laboratory tests.

The study duration will last for 12 weeks and patients will be monitored at week 0, week 1, week 2, week 4, week 8, and week 12 for 6 times. Urinary toxicology and visual analogue scales will be checked at each visit and laboratory chemistry at each visit.

Randomization

The study subjects will be randomly assigned by computer-generated numbers either to the lamotrigine or placebo group in a 1:1 ratio.

Dosage of trial medication

Trial medication and placebo will be sponsored by Lotus pharmaceutical, Taiwan. It is an extended release tablet form of lamotrigine or identical placebo. The preparation of double procedure will be handled by the Department of Pharmacy of Taipei City Hospital.

Once a subject enters the treatment phase (after randomization) the dosage of study medication will be 25 mg/before bed (or one half placebo tablet at night) for 7 days. On day 8 (visit 2 or the beginning of week 2), the dosage will be increased, as tolerated, to 50 mg/day for another week. After then, the dosage will be increased to 100 mg/day (QD and HS) for 2 weeks. After 4 weeks, the dosage may be kept or increased, as judged by investigator, at the range of 100mg to 200mg /day to the end of 12 weeks. The dosage may be decreased at any time because of side effects, but not less than 100 mg. If the patient prefers, he or she may take all of his or her daily dose of medication in the morning or evening.

The enroll period will be 2 years and total study duration will be 3 years.

Concomitant and prohibited medications

During study period, patients can take their original medications for systemic disorder. Due to patients with drug abuse usually have depressed mood, emotional disturbance or sleep problems during withdrawal period, benzodiazepines, or short acting novel hypnotics such as zolpidem or zaleplon can be used for ethical consideration. For those patient treated with antipsychotics due to drug-induced psychosis, the patients can be enrolled only when the psychotic symptoms remitted and lowest dose of antipsychotic can be used during the trial period. The prohibited medications include medications which have drug-drug interaction such as carbamazepine, phenytoin barbiturates, rifampicin, chlordiazepoxide and oral hypoglycaemics.

Primary endpoint

The primary endpoint will be the results from urinary drug screen of ketamine, and other substances including amphetamine, methylenedioxymethamphetamine, morphine and cannabis, which will be carried out at the baseline and during each visit of the study period.

Secondary endpoint

Subjective visual analogue scales of craving by patient and subjective clinical global impression of severity will be the second endpoint. The Brief Addiction Severity Index of ketamine use will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Current users of ketamine, including having a ketamine-positive urine
2. Meeting DSM-5 criteria for ketamine use disorder
3. Age between 18 to 65 years old
4. Women of childbearing age must have a negative pregnancy test to enroll in this study, agree to monthly pregnancy testing, and agree to use appropriate forms of birth control for the duration of the study.

Exclusion Criteria:

1. Significant medical conditions such as abnormal liver function or renal function confirmed by laboratory tests
2. Hypertension
3. A current cardiac condition or high risk of cardiovascular disease
4. Seizure disorders
5. Any another significant underlying medical condition which would contraindicate lamotrigine treatment
6. Meeting DSM-IV psychiatric classifications for schizophrenia, bipolar disorder, or other psychotic disorders
7. Meeting DSM-IV psychiatric classifications for substance use disorder other than ketamine within three month except tobacco or caffeine.
8. Exhibiting current suicidality or homicidality
9. Pregnant women, lactating women or women who are planning to be pregnant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09; Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Urine drug screen | 12 weeks
  Negative result of urinary drug toxicology screen of ketamine

SECONDARY OUTCOMES:
subjective visual analogue scales of craving | 12 weeks
  Scores of subjective visual analogue scales of craving rated by patient
Retention rate | 12 weeks
  Rate of patients stay in this trial

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Ku Lin, MD, Principal Investigator — Taipei City Hospital
Locations (1):
- Taipei City Hospital and Psychiatric Center, Taipei, Taiwan